CLINICAL TRIAL: NCT02959281
Title: The Application of Bio-impedance System NICAS and Hand-held Echocardiographic System (VSCAN) as Tools for Clinical Decision-making in the Treatment of In-patients With Cardio-renal Syndrome Type I
Brief Title: Bioimpedance and Hand-held Echocardiographay for Clinical Decision-making in Treatment of Cardio-renal Syndrome Type I
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollement failure
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Guy Dori, Head, Internal Medicine E, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMC-0081-16
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Cardio-Renal Syndrome
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodynamic data available (Experimental): Providing caring physicians with hemodynamic variables measured using the NICAS system.
  Interventions: Other: Providing caring physicians with hemodynamic variables
- Hemodynamic data not available (No Intervention): Hemodynamic variables measured using the NICAS system will not be provided to the caring physicians.

INTERVENTIONS:
Other: Providing caring physicians with hemodynamic variables — NICAS electrodes are applied to the skin of the forearm bilaterally (similar to EKG electrodes). Conductors, attached to the electrodes, connect the patient with the measuring system.
  Arms: Hemodynamic data available

SUMMARY:
The purpose of this study is to investigate whether hemodynamic data obtained by a noninvasive bio-impedance system (NICAS) sampled from patients with cardiorenal syndrome type I (CRS1) improve clinical outcomes. We hypothesize that hemodynamic data provided to the caring physician will improve management of CRS1 patients.

DETAILED DESCRIPTION:
Patients admitted to the hospital due to acute decompensation of heart failure (ADHF) may manifest some deterioration in their renal function. The latter is associated with unfavorable outcomes: prolonged hospitalization and death. Cardiorenal syndrome type 1 (CRS1) is defined as a deterioration in renal function manifested by an increase in serum creatinine level by >0.3 mg% compared to patient's baseline level. The etiology of CRS1 is not clear and may be related to body fluid overload congesting the kidneys or dehydration reducing perfusion to the kidneys. Body fluid status is affected by diuretics. Presently, the practitioner has no objective data to assess whether CRS1 resulted from fluid overload or dehydration.

In this study investigators plan to measure hemodynamic parameters from all patients admitted with CRS1 to our department. Parameters will be measured using the noninvasive bio-impedance system (NICAS). Randomly, patients will be allocated to either a study or control group. In the study group, the hemodynamic variables of the NICAS system will be available to the caring physicians. The physicians will use the data according to their discretion. The hemodynamic system is a decision making supporting system and therefore the physician may use the data according to his/her understanding. In the control group, the hemodynamic variables of the NICAS system will not be available to the caring physicians.

We hypothesize that using the NICAS system as a decision making supporting system will improve patient management by decreasing length of hospitalization, and shortening the time interval to reverse creatinine to its baseline level.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for acute decompensation of heart failure and developed cardiorenal syndrome (all three criteria below are required):

A. Evidence of heart failure defined by either (i) or (ii) and (iii), where:

(i) is clinical complaints of dyspnea or leg swelling or fatigue (ii) is clinical findings of pulmonary rales, leg edema, or congestion on chest film (iii) is recent (within 1 year of admission) echocardiographic examination demonstrating heart failure B. Patient as in A (above) whos serum creatinine level on admission is 0.3 mg% greater than patient's baseline.

C. Patient capable of submitting informed consent

Exclusion Criteria:

* Other causes for dyspnea or leg edema (e.g. exacerbation of COPD, pneumonia, liver cirrhosis, hypoalbuminemia, nephrotic syndrome)
* other causes for acute renal failure (e.g. contrast media nephropathy 10 days prior to admission, use of NSAIDS or antibiotics (aminoglycosides, quinolones), diarrhea, vomiting, rhabdomyolysis, seizures, sepsis.
* Anemia (Hb<8 gr%)
* significant bleeding (upper or lower GI, hemoptysis)
* BMI>40, or BMI<18
* Signs of a new myocardial infarction by EKG, and increase in troponin levels to levels 1.5 above baseline levels.
* Hypothyroidism
* Addison's disease
* patient on Hemo- or peritoneal dialysis
* Mechanical ventillation

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-16 (Actual)

PRIMARY OUTCOMES:
Mean hospitalization duration (in days) | 2 months
  Time of hospitalization is defined from time of recruitment till the time patient is ready for discharge.

SECONDARY OUTCOMES:
Time from maximum serum creatinine level to patient's discharge | 2 months
  Time from maximum serum creatinine level to time when patient is ready for discharge
Maximum difference in serum creatinine level | 2 months
  This outcome is defined by the maximum serum creatinine level obtained during the followup of the patient minus patient's mean serum creatinine level

CONTACTS AND LOCATIONS:
Overall Officials: Guy Dori, MD, DSc, Principal Investigator — haemek medical center

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to share the IPD with any body. After completion of study we plan to publish results.

REFERENCES:
- [Background] Ronco C, Cicoira M, McCullough PA. Cardiorenal syndrome type 1: pathophysiological crosstalk leading to combined heart and kidney dysfunction in the setting of acutely decompensated heart failure. J Am Coll Cardiol. 2012 Sep 18;60(12):1031-42. doi: 10.1016/j.jacc.2012.01.077. Epub 2012 Jul 25. PMID 22840531